CLINICAL TRIAL: NCT02400034
Title: A Randomized Controlled Trial Comparing Force of Stream to Traditional Retrograde Fill Voiding Trial After Midurethral Sling With or Without Vaginal Prolapse Surgery
Brief Title: Comparing Voiding Trials After Midurethral Sling for Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Harvey Winkler, FPMRS Fellowship Director, Co-Chair Division of Urogynecology, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-667
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Stress Urinary Incontinence; Urethral Hypermobility; Cystocele
Keywords: midurethral sling; Voiding trial; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Cystocele | interventions — Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FAST voiding trial method (Active Comparator): 1) Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water. 2) catheter is removed; 3) Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). 4) The patient will subjectively quantify their FOS via VAS scale. 5) If VAS scale >50 (=50%) the catheter will remain out, patient is discharged home without measuring a PVR 6) If VAS scale is from 0-49 (= 0-49%) a PVR will be checked via bladder scan. If PVR is <500 the patient will be discharged WITHOUT a catheter; If PVR is >500 the patient will be discharged WITH a catheter. If she is discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days
  Interventions: Other: Voiding trial
- Retrograde fill voiding trial method (Active Comparator): 1) Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water. 2) catheter is removed; 3) Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). 4) The patient will subjectively quantify their FOS via VAS scale (however this information will only be used for research purposes). 5) If she voids >/= 2/3 (200cc) the catheter will remain out as she will have passed her voiding trial. If she voids < 200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial in 2-5 days.
  Interventions: Other: Voiding trial

INTERVENTIONS:
Other: Voiding trial — 1 of 2 tests to assess bladder function after midurethral sling surgery with and without anterior or posterior colporrhaphy
  Other Names: voiding

SUMMARY:
Urinary incontinence is a prevalent health and quality of life concern affecting almost half of women over the age of 20. Urinary retention (abnormal holding of urine) is a concern of many surgeons who perform midurethral sling surgery. All patients after outpatient midurethral sling or vaginal prolpase surgery must complete a voiding trial if they are to be discharged without a catheter. The purpose of this study is to compare two different types of postoperative voiding trials to determine which leads to less post-operative issues, such as urinary retention requiring catheterization. You are being asked to participate because you are having midurethral sling surgery, either with or without vaginal prolapse repair.

DETAILED DESCRIPTION:
Urinary incontinence is a prevalent health and quality of life concern affecting an estimated 49.6% of women over the age of 20 years in the USA. (1) Of these, 49.8% describe pure stress urinary incontinence (SUI) and 34.3% report mixed stress and urgency urinary incontinence. (1)

Midurethral sling (MUS) surgery is used to treat women with SUI, but accepted protocols for voiding trials after midurethral sling placement do not exist. Primarily, many surgeons measure postvoid residual (PVR) urine volume. This is done by retrograde filling of the bladder with a predetermined amount of normal saline or water. The catheter is then removed and the patient is permitted to void into a collection basin. The amount in the basin is subtracted from the filled amount. The need for catheterization is generally based on arbitrarily determined ratios of voided urine to PVR or postoperative.

The acceptable amount voided during catheterization varies among practitioners. In a study by Kleeman et al, the patient was required to void >50% of volume filled during retrograde fill for discharge from hospital without an indwelling Foley catheter (2). Pulvino et al, required that the patient void > 2/3 the amount of the volume placed during retrograde fill (3). The force of stream trial (FAST) does not prioritize amount voided, but rather the patient's subjective force of stream. The bladder is retrograde filled with 300cc normal saline or water and the patient is instructed to void.. Using FAST, a patient uses a VAS scale to quantify her force of stream. If she states that her Force of Stream (FOS) is >50% stronger than prior to surgery, independent of the amount voided, she is discharged without a catheter. If the FOS is <50% a PVR via bladder scan is performed. If her PVR is <500cc the patient was discharged home without a catheter in place. If the PVR, via bladder scan was > 500cc she was discharged with a catheter. Ingber et. Al. showed the FAST method was a safe method for predicting postoperative voiding dysfunction and/or urinary retention. No patients presented to the office or emergency room for voiding dysfunction or urinary retention (4).

Urinary retention is a concern of many surgeons who perform midurethral sling surgery; 25% of urologists routinely discharge patients home with a catheter and 31% admit patients overnight or for 23 hour observation, with 42% doing so for the primary purpose of facilitating the voiding trial. (5)

Published catheterization rates for these protocols can approach 39%. (6,7) Temporary catheterization does not pose a significant medical risk, but it is perceived as an inconvenience and source of discomfort for many patients. Proper care of an indwelling foley catheter requires extra teaching from nursing and/or house staff.

No randomized control trials (RCT) have been performed comparing the FAST method to the traditional retrograde voiding trial. In our practice we assess postoperative voiding function using the retrograde fill with 300cc saline or water. We also require a 2/3 quantity voided for discontinuation of catheter.

All patients after outpatient midurethral sling or vaginal prolpase surgery must complete a voiding trial if they are to be discharged without a catheter. This is standard of care and followed in our practice. We would like to compare both postoperative voiding trials in patients who have undergone surgical repair concomitant midurethral sling with or without anterior colporrhaphy. We will include those patients who also had an anterior colporrhaphy at time of sling placement as this procedure is commonly performed at the time of sling placement for stablization of MUS. We will assess the number of emergent or unexpected visits for voiding dysfunction. An unexpected visit to the office will be defined as any visit outside of the patient's prior scheduled postoperative visits.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative patients after placement of midurethral sling (retropubic sling or transobturator) with or without anterior or posterior colporrhaphy.
2. Ability to provide informed consent and complete all study requirements

Exclusion Criteria:

1. Patients who underwent a surgery that requires long term catheterization (i.e fistula repair or urethral diverticulum)
2. Patients who sustained a cystotomy during surgery as our divisional protocol is to send these patients home with a Foley catheter for 5-14 days without a voiding trial
3. Patients who had an apical repair for pelvic organ prolapse (Uterosacral vaginal vault suspension, Abdominal sacral colpopexy, sacrospinous ligament fixation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of emergency room visits or unexpected visits to the office within 6 weeks postoperatively for voiding dysfunction or suspected infection | 6 weeks
  Any additional visit outside the patient's scheduled postoperative visits to the emergency room, urgent care facility or doctor's office will be recorded for up to 6 six weeks postoperatively

SECONDARY OUTCOMES:
Number of patients sent home with a catheter | 6 weeks
  the number of patients in each arm who are sent home with a catheter will be recorded
Number of patients with reported UTI | 6 weeks
Time to discharge from hospital | 6 weeks
  Time upon arrival to Post Anesthesia Care Unit to discharge to home will be calculated for each arm
Patient satisfaction with postoperative bladder function | 6 weeks
  American Urological Association Symptom Score (AUASS); Urinary Distress Inventory (UDI-6)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey A Winkler, MD, Principal Investigator — North Shore LIJ Divsion of Female Pelvic Medicine and Reconstructive Surgery
Locations (1):
- Urogynecology, Female Pelvic Medicine and Reconstructive Surgery, Great Neck, New York, United States

REFERENCES:
- [Background] Stav K, Dwyer PL, Rosamilia A, Schierlitz L, Lim YN, Chao F, De Souza A, Thomas E, Murray C, Conway C, Lee J. Repeat synthetic mid urethral sling procedure for women with recurrent stress urinary incontinence. J Urol. 2010 Jan;183(1):241-6. doi: 10.1016/j.juro.2009.08.111. PMID 19913831
- [Background] Kleeman S, Goldwasser S, Vassallo B, Karram M. Predicting postoperative voiding efficiency after operation for incontinence and prolapse. Am J Obstet Gynecol. 2002 Jul;187(1):49-52. doi: 10.1067/mob.2002.124841. PMID 12114887
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Ingber MS, Vasavada SP, Moore CK, Rackley RR, Firoozi F, Goldman HB. Force of stream after sling therapy: safety and efficacy of rapid discharge care pathway based on subjective patient report. J Urol. 2011 Mar;185(3):993-7. doi: 10.1016/j.juro.2010.10.050. Epub 2011 Jan 19. PMID 21247598
- [Background] Barron KI, Savageau JA, Young SB, Labin LC, Morse AN. Prediction of successful voiding immediately after outpatient mid-urethral sling. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Nov;17(6):570-5. doi: 10.1007/s00192-005-0064-8. Epub 2006 Apr 1. PMID 16583182
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Peleg AY, Hooper DC. Hospital-acquired infections due to gram-negative bacteria. N Engl J Med. 2010 May 13;362(19):1804-13. doi: 10.1056/NEJMra0904124. No abstract available. PMID 20463340
- [Background] El-Barky E, El-Shazly A, El-Wahab OA, Kehinde EO, Al-Hunayan A, Al-Awadi KA. Tension free vaginal tape versus Burch colposuspension for treatment of female stress urinary incontinence. Int Urol Nephrol. 2005;37(2):277-81. doi: 10.1007/s11255-004-6101-6. PMID 16142556
- [Background] Barber MD, Kleeman S, Karram MM, Paraiso MF, Walters MD, Vasavada S, Ellerkmann M. Transobturator tape compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):611-21. doi: 10.1097/AOG.0b013e318162f22e. PMID 18310363
- [Background] Ward KL, Hilton P; UK and Ireland TVT Trial Group. Tension-free vaginal tape versus colposuspension for primary urodynamic stress incontinence: 5-year follow up. BJOG. 2008 Jan;115(2):226-33. doi: 10.1111/j.1471-0528.2007.01548.x. Epub 2007 Oct 25. PMID 17970791
- [Background] Liapis A, Bakas P, Creatsas G. Long-term efficacy of tension-free vaginal tape in the management of stress urinary incontinence in women: efficacy at 5- and 7-year follow-up. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Nov;19(11):1509-12. doi: 10.1007/s00192-008-0664-1. Epub 2008 Jun 10. PMID 18542836